CLINICAL TRIAL: NCT02596360
Title: Dextromethorphan Effect on Central Sensitization to Pain in Healthy Volunteers
Acronym: Hydex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0248; 2015-003271-30 (Registry Identifier: 2015-003271-30)
Record Dates: First submitted 2015-10-19; First posted 2015-11-04 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Experimental Pain; Hyperalgesia
Keywords: Antinociception; Freeze-induced hyperalgesia model; Dextromethorphan; NMDA-receptors; Pharmacogenetic; CYP3A4 gene; MDR1 gene
MeSH Terms: conditions — Hyperalgesia | interventions — Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dextromethorphan (Experimental): The study design is divided in two study sequences and each subject participates in the two study sequences and receive the two treatments (dextromethorphan and placebo).
  Interventions: Drug: Pulmodexane® 30mg
- Placebo (Placebo Comparator): The study design is divided in two study sequences and each subject participates in the two study sequences and receive the two treatments (dextromethorphan and placebo).
  Interventions: Drug: lactose

INTERVENTIONS:
Drug: Pulmodexane® 30mg — The study design is divided in two study sequences and each subject participates in the two study sequences and receive the two treatments (dextromethorphan and placebo).
  Arms: Dextromethorphan
Drug: lactose — The study design is divided in two study sequences and each subject participates in the two study sequences and receive the two treatments (dextromethorphan and placebo).
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the anti-hyperalgesic effect of dextromethorphan in healthy volunteers compared to placebo.

DETAILED DESCRIPTION:
This is a cross-over group, double-blind, randomized clinical trial in healthy volunteers comparing dextromethorphan and inactive control on freeze-induced hyperalgesia, experimental pain, diffuse noxious inhibitory control (DNIC), pupillary reaction and reaction time.

The influence of CYP3A4 and MDR1 polymorphism on the dextromethorphan analgesic efficacy will be measured.

The study design is divided in two study sequences and each subject participates in the two study sequences and receive the two treatments (dextromethorphan and placebo).

Each study sequence consists of 3 assessment days (Day -1, Day 0 = first treatment administration and Day 1).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Aged between 18 and 45 years
* CYP2D6 Extensive and Intermediate metabolizers
* Body mass index (BMI) between 19 and 30 kg/m2
* Systolic blood pressure between 100 and 150 mmHg, diastolic blood pressure between 50 and 90 mmHg, heart rate between 45 and 90 beats per minute
* Without treatment during the 7 days before inclusion specially no use of analgesic and anti-inflammatory drugs
* Cooperation and understanding enough to conform to the study obligations
* Having given free informed written consent
* Affiliated to the French Social Security
* Inscription or acceptation of inscription in the national register of volunteers involved in trials.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Lactose intolerance
* Hypertension
* History of stroke
* Severe heart failure
* Severe hepatic impairment
* Shortness of breath
* Congenital galactosemia, glucose-galactose malabsorption, lactase deficiency
* Association with linezolid
* Pre-existence or history of peripheral neuropathy due to a cause different from neurotoxic chemotherapy
* Diabetes (type I and II)
* CYP2D6 Poor and Ultra-rapid metabolizers
* AST, ALT, total bilirubin twice the average
* Dextromethorphan intake during the 7 days before inclusion
* Medical and surgical history incompatible with the study
* Disease progression during inclusion
* Excessive consumption of alcohol (> 50g/day), tobacco (≥ 10 cigarettes/day), coffee, tea or drinks with caffeine (equivalent to more than 4 cups a day) or any addiction to drugs
* Subject lacking concentration during tests training and low test results reproducibility
* Subject does not meet the selection criteria for its ability to discriminate sensations to noxious stimuli during psychometric tests
* Subject exclusion period, or the total allowable compensation exceeded
* Subject undergoing a measure of legal protection (guardianship, supervision

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of percentage changes in mechanical pain thresholds (MPT) using electronic von frey in secondary hyperalgesic zone (Z2) | at Day 0 after treatment administration: 1 hour post-dose (T0+1h), 2 hours post-dose (T0+2h) and 3 hours post-dose (T0+3h).

SECONDARY OUTCOMES:
Area under the curve (AUC) of percentage changes in mechanical pain thresholds (MPT) using electronic von frey in control skin zone (Z0) and primary hyperalgesic zone (Z1) | at D0 T0+1h, T0+2h and T0+3h after treatment administration
Percentage changes in mechanical pain thresholds (MPT) using electronic von frey in control skin zone (Z0) | at Day 0 after treatment administration: 1 hour post-dose (T0+1h), 2 hours post-dose (T0+2h) and 3 hours post-dose (T0+3h).
Percentage changes in mechanical pain thresholds (MPT) using electronic von frey in primary hyperalgesic zone (Z1) | at Day 0 30 min before treatment (T0-30min ) and at Day 0 after treatment administration: 1 hour post-dose (T0+1h), 2 hours post-dose (T0+2h) and 3 hours post-dose (T0+3h) and at Day 1 after treatment administration: 24,5 hours post-dose (T0+24h30).
Conditioned Pain Modulation (CPM) assessment | at Day -1 before treatment and Day 0 30 min before treatment (T0-30min)
Reaction time assessment using RTI CANTAB® test | at Day -1 before treatment and Day 0 30 min before treatment (T0-30min), after treatment administration: 1 hour post-dose (T0+1h) and 3 hours post-dose (T0+3h) and at Day 1 after treatment administration: 24,5 hours post-dose (T0+24h30).
Determination of potential central effects of dextromethorphan measuring pupillary reaction | at Day 0 30 min before treatment (T0-30min ) and at Day 0 after treatment administration: 1 hour post-dose (T0+1h), 2 hours post-dose (T0+2h) and 3 hours post-dose (T0+3h) and at Day 1 after treatment administration: 24,5 hours post-dose (T0+24h30).
  Determination of potential central effects of dextromethorphan measuring pupillary reaction assessing the diameter of the pupil in real time in scotopic conditions (e.g. size variation [mm]; contraction speed [mm.s-1]; contraction latency [ms]) at Day 0 30 min before treatment (T0-30min ) and at Day 0 after treatment administration: 1 hour post-dose (T0+1h), 2 hours post-dose (T0+2h) and 3 hours post-dose (T0+3h) and at Day 1 after treatment administration: 24,5 hours post-dose (T0+24h30).
  - Study of genetic polymorphism of cytochrome P450 3A4 and MDR1 gene through study completion, up to 6 months.
Study of genetic polymorphism of cytochrome P450 3A4 and genetic polymorphism of MDR1 gene | up to 6 months.
Dosage of plasma concentration of dextromethorphan and dextromethorphan's metabolites from blood collections | at Day 0 30 min before treatment (T0-30min ) and at Day 0 after treatment administration: 2 hours post-dose (T0+2h) and at Day 1 after treatment administration: 24,5 hours post-dose (T0+24h30).

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France